CLINICAL TRIAL: NCT00143286
Title: A 52-Week Multicenter Study Evaluating the Safety and Efficacy of Varenicline ( CP-526,555) for the Maintenance of Smoking Cessation
Brief Title: A 52-Week Multicenter Study Evaluating the Safety and Efficacy of Varenicline for the Maintenance of Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051035
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline (CP-526,555)

SUMMARY:
The primary purpose of this study is a comparison of abstinence maintenance in subjects randomized to double-blind varenicline or placebo from Weeks 13 -24 in subjects who responded to an intial 12-week open label course of varenicline, with post-treatment follow-up of smoking status to Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Subjects with clinically significant cardiovascular disease in the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2003-04; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence Weeks 13 -24.

SECONDARY OUTCOMES:
Continuous abstinence Weeks 13-52
Long term quit rate at Week 52
7-day Point Prevalence of abstinence at Weeks 24, 52
4-week Point Prevalence of abstinence at Week 52
Time to first cigarette post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (6):
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Mogadore, Ohio
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Canada (6):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Cornwall, Prince Edward Island
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Pfizer Investigational Site, Prague, Czechia
- Denmark (3):
  - Pfizer Investigational Site, Hellerup, Copenhagen
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Frederikssund
- Norway (3):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Hønefoss
  - Pfizer Investigational Site, Oslo
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Stockholm
- United Kingdom (2):
  - Pfizer Investigational Site, London, Surrey
  - Pfizer Investigational Site, London

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hajek P, Tonnesen P, Arteaga C, Russ C, Tonstad S. Varenicline in prevention of relapse to smoking: effect of quit pattern on response to extended treatment. Addiction. 2009 Sep;104(9):1597-602. doi: 10.1111/j.1360-0443.2009.02646.x. PMID 19686530
- [Derived] Tonstad S, Tonnesen P, Hajek P, Williams KE, Billing CB, Reeves KR; Varenicline Phase 3 Study Group. Effect of maintenance therapy with varenicline on smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):64-71. doi: 10.1001/jama.296.1.64. PMID 16820548
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051035&StudyName=A+52%2DWeek+Multicenter+Study+Evaluating+the+Safety+and+Efficacy+of+Varenicline+for+the+Maintenance+of+Smoking+Cessation